CLINICAL TRIAL: NCT06707519
Title: A Prospective, Single Center Study to Test the Validity and Feasibility of Circulating Tumor DNA in Blood, Sputum and Alveolar Fluid, as Well as Exhaled Volatile Organic Compounds as Biomarkers in Non-Small Cell Lung Cancer
Brief Title: NSCLC Liquid Biopsies and Exhaled VOC
Status: Recruiting | Type: Observational
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Yaron Shargall, Professor, St. Joseph's Healthcare Hamilton
Other Study IDs: 14065
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer; Circulating Tumor DNA
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study is to determine the feasibility of recruiting participants and using sputum, Bronchoalveolar lavage (BAL) and exhaled Volatile Organic Compounds (VOC) in addition to blood, as biological samples for detecting mutations in extracted cell-free DNA in non-small cell lung cancer (NSCLC) patients, before and after surgery, and any recurrence within a 24-month postoperative follow-up period.

This is a pilot feasibility study, proposed as a 24-month prospective, single-center, non-interventional, observational trial with NSCLC-adenocarcinoma patients indicated for resection surgery with curative intent.

DETAILED DESCRIPTION:
Circulating tumor DNA (ctDNA) is increased in patients with lung cancer, and may allow detecting minimal residual disease and disease recurrence, preceding radiological detection. Detecting ctDNA in bronchoalveolar lavage/Sputum was never validated and may offer advantages over blood ctDNA, and serve as a novel biomarker for lung cancer surveillance. Lung cancer detection is possible with eNose systems with a high negative predictive value and allows prediction of treatment response to PD1 inhibitors, monitoring response to PD1 inhibitors and predicting the presence of EGFR mutations. it is reasonable to anticipate exhaled VOC to aid in detection of cancer recurrence.

The study propulsion is patients undergoing surgical resection with curative intent for NSCLC, adenocarcinoma subtype at St. Joseph's Healthcare Hamilton and the Firestone Institute of Respiratory Health , above 18 years, able to provide consent. The study procedure is collecting blood, sputum, BAL samples, exhaled VOC will be collected at the following time-points/visits: (i) Visit 1 (V1): pre surgical resection; (ii) V2: immediately before discharge from hospital post-resection; (iii) V3,4,5 : 6, 12, 24 months post-surgery; (iv) V6: unscheduled at any sign of recurrence. to note, blood sputum and BAL will be collected at visit 1 and 2 from everyone and at visits 3-6 only from those who harbor a mutation of interest.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age
* Patient must be able to provide consent
* Patients undergoing surgical resection with curative intent for non-small cell lung cancer at St. Joseph's Healthcare Hamilton and Firestone Institute for Respiratory Health.

Exclusion Criteria:

* Resection done with non-curative intent or metastatic disease
* other malignancies
* Patients with previously treated malignancy less than 5 years prior to current resection (not including skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical resection with curative intent for NSCLC, adenocarcinoma subtype at St. Joseph's Healthcare Hamilton and the Firestone Institute of Respiratory Health , above 18 years, able to provide consent
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | December 2025
  the proportion of eligible participants recruited (threshold >75%)
Data completion rate | December 2025
  proportion of samples that are usable (threshold >80%)
Safety, adverse events | December 2025
  any adverse events (threshold <10%)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
There is currently no decision on whether the IPD will be available to other researchers.